CLINICAL TRIAL: NCT07041840
Title: ReModeling in ST-elevation myocARrdial Infarction: a Comparison of Left VEntricuLar Functions in Long-term Follow-up Among STEMI Patients: The MARVEL Study
Brief Title: ReModeling in ST-elevation myocARrdial Infarction: a Comparison of Left VEntricuLar Functions in Long-term Follow-up Among STEMI Patients
Acronym: MARVEL
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Mattia Alberti, Dr, University of Pisa
Other Study IDs: MARVEL
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI: STEMI

SUMMARY:
Patients diagnosed with STEMI who underwent pPCI were included in this study. The investigators collected comprehensive data on each patient's status, including laboratory findings such as NT-proBNP, troponin levels, and inflammatory profile assessed by leukocyte count, C-reactive protein, interleukin-1, and interleukin-6. Additionally, electrocardiographic and echocardiographic features, details of the coronary intervention procedure, hospital stay duration, complications, and medical treatments were recorded.

Comprehensive transthoracic echocardiograms (TTE) were performed at admission and before discharge. Myocardial tissue characterization was conducted by cardiac magnetic resonance (CMR) imaging before discharge, assessing intramyocardial hemorrhage (IMH), microvascular obstruction (MVO), infarct size (IS), area at risk (AAR), salvaged myocardium, and salvage index.

At the six-month follow-up, laboratory tests, CMR imaging, and TTE were repeated, along with a thorough clinical evaluation. LVR was defined by one of the following criteria: a 20% increase in end-diastolic volume by TTE or 12% by CMR, a 15% increase in end-systolic volume, a sphericity index greater than 42% (CMR only), the emergence of new concentric hypertrophy, or a reduction greater than 10% in left ventricular ejection fraction (LVEF).

DETAILED DESCRIPTION:
Patients diagnosed with STEMI who underwent pPCI were included in this study. The investigators collected comprehensive data on each patient's status, including laboratory findings such as NT-proBNP, troponin levels, and inflammatory profile assessed by leukocyte count, C-reactive protein, interleukin-1, and interleukin-6. Additionally, electrocardiographic and echocardiographic features, details of the coronary intervention procedure, hospital stay duration, complications, and medical treatments were recorded.

Comprehensive transthoracic echocardiograms (TTE) were performed at admission and before discharge. Myocardial tissue characterization was conducted by cardiac magnetic resonance (CMR) imaging before discharge, assessing intramyocardial hemorrhage (IMH), microvascular obstruction (MVO), infarct size (IS), area at risk (AAR), salvaged myocardium, and salvage index.

At the six-month follow-up, laboratory tests, CMR imaging, and TTE were repeated, along with a thorough clinical evaluation. LVR was defined by one of the following criteria: a 20% increase in end-diastolic volume by TTE or 12% by CMR, a 15% increase in end-systolic volume, a sphericity index greater than 42% (CMR only), the emergence of new concentric hypertrophy, or a reduction greater than 10% in left ventricular ejection fraction (LVEF).

ELIGIBILITY:
Inclusion Criteria:

* STEMI

Exclusion Criteria:

* Contraindication to CMR imaging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Remodeling | 36 months
  Left Ventricular Remodeling was defined by one of the following criteria: a 20% increase in end-diastolic volume by Trans-Thoracic Echocardiography or 12% by Cardiac Magnetic Resonance (CMR) Imaging, a 15% increase in end-systolic volume, a sphericity index greater than 42% (CMR only), the emergence of new concentric hypertrophy, or a reduction greater than 10% in left ventricular ejection fraction (LVEF).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Cisanello Hospital, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request